CLINICAL TRIAL: NCT06129422
Title: A Phase I Trial to Assess Safety, Tolerability, Pharmacokinetics, Radiation Dosimetry, and Positron Emission Tomography (PET) Imaging Properties of 89Zr-labeled hNd2 (NMK89) in Patients With Pancreatic Cancer Histologically Positive for MUC5AC
Brief Title: Safety, Tolerability, Pharmacokinetics, Radiation Dosimetry, and PET Imaging Properties of 89Zr-labeled hNd2 (NMK89) in Patients With Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nihon Medi-Physics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NMK89P101
Record Dates: First submitted 2023-10-27; First posted 2023-11-13 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer; MUC5AC
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NMK89 (Experimental): Patients will receive a single infusion of NMK89
  Interventions: Drug: NMK89

INTERVENTIONS:
Drug: NMK89 — Route of administration: intravenous infusion

SUMMARY:
This trial will be a non-randomized, Phase I trial to evaluate safety, tolerability, biodistribution, radiation dosimetry, pharmacokinetics and PET imaging properties following an infusion of 37 MBq (1 mCi) of 89Zr-labeled hNd2* (NMK89) in patients with pancreatic cancer that are positive for MUC5AC. Image acquisition is conducted using a PET/CT machine.

* hNd2: Recombinant humanized Nd2 (anti-human MUC5AC monoclonal antibody)

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent.
2. Male or female ≥ 18 years of age.
3. Histologically confirmed diagnosis of pancreatic adenocarcinoma.
4. Willing to provide biopsy specimens for purposes of confirmation of MUC5AC expression.
5. Confirmed MUC5AC expression at pre-screening.
6. Measurable disease.
7. Female patients of child-bearing potential must have a negative serum pregnancy test within 30 days prior to infusion of NMK89.
8. Willing to comply with the study protocol requirements.
9. Willing to provide a tumor resection specimen or biopsy specimen, if the patient undergoes tumor resection or biopsy between Day 16 and Day 60.

Exclusion Criteria:

1. Known hypersensitivity to the investigational medicinal product (IMP) or any of the excipients.
2. History of another primary cancer within the 2 years prior to enrollment, except for the curatively treated in situ cancers.
3. Exposure to any investigational treatments within 30 days prior to the planned date of infusion of NMK89.
4. Ongoing toxicity ≥ Grade 2.
5. Pleural effusion or peritoneal fluid ≥ Grade 3.
6. Active hepatitis B, hepatitis C, HIV, or other progressing infectious disease.
7. Uncontrolled diabetes.
8. Autoimmune disease or idiopathic thrombocytopenic purpura.
9. Exposure to any radiopharmaceuticals.
10. Planned antineoplastic therapies on the planned date of NMK89 infusion.
11. Use of bevacizumab or any other anti-angiogenic agent.
12. Uncontrolled intercurrent illness.
13. ECOG PS: ≥ 2.
14. Participants do not have adequate organ and marrow function.
15. Female patients that are pregnant or breast-feeding.
16. Positive urine screen for illegal drugs, or abuse of prescribed drugs at Screening.
17. Participants with contraindications to contrast agent injection used for diagnostic CT.
18. Deemed inappropriate to participate by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-10-31 (Actual); Primary Completion 2025-10-07 (Actual); Study Completion 2025-10-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of a single infusion of NMK89: physical examination 1 | Screening to Day 8
  Body weight
Safety and tolerability of a single infusion of NMK89: physical examination 2 | Screening
  Height
Safety and tolerability of a single infusion of NMK89: vital sign 1 | Screening to Day 8
  Body temperature
Safety and tolerability of a single infusion of NMK89: vital sign 2 | Screening to Day 8
  Heart rate
Safety and tolerability of a single infusion of NMK89: vital sign 3 | Screening to Day 8
  Systolic blood pressure (SBP)
Safety and tolerability of a single infusion of NMK89: vital sign 4 | Screening to Day 8
  Diastolic blood pressure (DBP)
Safety and tolerability of a single infusion of NMK89: 12-lead ECG (Electrocardiogram) 1 | Screening to Day 8
  PR interval
Safety and tolerability of a single infusion of NMK89: 12-lead ECG 2 | Screening to Day 8
  RR interval
Safety and tolerability of a single infusion of NMK89: 12-lead ECG 3 | Screening to Day 8
  QRS interval
Safety and tolerability of a single infusion of NMK89: 12-lead ECG 4 | Screening to Day 8
  QT
Safety and tolerability of a single infusion of NMK89: 12-lead ECG 5 | Screening to Day 8
  Corrected QT
Safety and tolerability of a single infusion of NMK89: Frequency and severity of abnormal adverse events (AEs) (National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v 5.0)) | Baseline up to Day 60
Safety and tolerability of a single infusion of NMK89: Clinical laboratory finding - hematology | Screening to Day 8
  Hematology included hemoglobin, hematocrit, mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), white blood cell count (total and differential: leukocytes, neutrophils, eosinophils, basophils, lymphocytes, monocytes), red blood cells, platelets.
Safety and tolerability of a single infusion of NMK89: Clinical laboratory finding - serum chemistry | Screening to Day 8
  Serum chemistry included sodium, potassium, chloride, calcium, glucose, creatinine, urea or BUN, albumin, total bilirubin, aspartate transaminase (AST), alanine transaminase (ALT), alkaline phosphatase, gamma-glutamyl transferase (GGT), lipase, amylase and total protein.
Safety and tolerability of a single infusion of NMK89: Clinical laboratory finding - clotting factors | Screening to Day 8
  Clotting factors included prothrombin time (quick), reagent-independent prothrombin ratio (international normalized ratio; INR), activated partial thromboplastin time (aPTT).
Safety and tolerability of a single infusion of NMK89: Clinical laboratory finding - urinalysis | Screening to Day 8
  Urinalysis included specific gravity, pH, protein, glucose, blood, leukocytes, ketones, nitrite, albumin, creatinine.
Safety and tolerability of a single infusion of NMK89: Frequency and severity of abnormal ECOG PS (Eastern Cooperative Oncology Group Performance Status) | Screening to Day 8

SECONDARY OUTCOMES:
Biodistribution: Fractional injected 89Zr radioactivity values (percentage of injected dose(%ID)) | Day 1 to Day 8
  PET/CT image acquisitions will be obtained to assess biodistribution of NMK89 in normal tissues and tumors in patients.
Biodistribution: Time-integrated activity coefficients (TIACs) (hr) | Day 1 to Day 8
  PET/CT image acquisitions will be obtained to assess biodistribution of NMK89 in normal tissues and tumors in patients.
Radiation Dosimetry of NMK89: Normalized radiation absorbed doses and normalized effective dose | Day 1 to Day 8
  Whole-body radiation dosimetry of NMK89 in patients will be estimated.
Optimization of positron emission tomography (PET) Scan Protocol: Optimal time from injection to start of PET | Day 1 to Day 8
  Optimal time from injection to start of PET acquisition will be determined.
Predictive radiation dosimetry of hNd2 labeled with therapeutic radionuclide: Normalized absorbed doses and normalized effective dose | Day 1 to Day 8
  Whole-body radiation dosimetry (if hNd2 will be labeled with a therapeutic radionuclide) will be estimated.
Blood Pharmacokinetics (PK): Concentration of total antibody in blood | Pre-infusion (baseline) to Day 8
  PK will be evaluated based on concentration of total antibody obtained within defined volumes of blood.
Blood Pharmacokinetics (PK): Concentration of total radioactive counts in blood | Day 1 to Day 8
  PK will be evaluated based on concentration of total radioactive counts obtained within defined volumes of blood.
Blood Pharmacokinetics (PK): Abundance ratio of unmetabolized 89Zr-labeled hNd2(%) | Day 1 to Day 8
  To calculate this ratio, the count of metabolites and non-metabolic components is obtained
Urine Pharmacokinetics (PK): Concentration of total antibody in urine | Pre-infusion (baseline) to Day 8
  PK will be evaluated based on concentration of total antibody obtained within defined volumes of urine.
Urine Pharmacokinetics (PK): Concentration of total radioactive counts in urine | Day 1 to Day 8
  PK will be evaluated based on concentration of total radioactive counts obtained within defined volumes of urine.
Urine Pharmacokinetics (PK): Radioactivity counts of 89Zr-labeled hNd2 and metabolites components | Day 1 to Day 8
  Radioactivity counts of 89Zr-labeled hNd2 and metabolites components are measured by magnetic separation, and the abundance ratio of unmetabolized 89Zr-labeled hNd2 (%) will be calculated.
Biological half-life of the radionuclide (hr) | Day 1 to Day 8
  Biological half-life of the radionuclide (hr) will also be estimated.
Public Safety: Radiation measurement | Day 1
  Public safety will be assessed by acquiring dosimeter readings of a patient following infusion.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Moffitt Cancer Center, Tampa, Florida
  - BAMF Health, Grand Rapids, Michigan
  - Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nakata N, Kobashi N, Okumura Y, Sato M, Matono M, Otsuki K, Tanaka A, Hayashi A. Radiation dosimetry and efficacy of an 89Zr/225Ac-labeled humanized anti-MUC5AC antibody. Nucl Med Biol. 2022 May-Jun;108-109:33-43. doi: 10.1016/j.nucmedbio.2022.02.003. Epub 2022 Feb 26. PMID 35276446
- [Background] Kulkarni HR, Maupin KA, Brennan T, Forsberg J, Rogers D, Olson M, Mancini BR, Chang A, Chandana SR, Kobayashi R. First-in-Human Total-Body PET/CT Imaging Using 89Zr-Labeled MUC5AC Antibody in a Patient with Pancreatic Adenocarcinoma. J Nucl Med. 2024 Nov 1;65(11):1815. doi: 10.2967/jnumed.124.268074. No abstract available. PMID 39237345